CLINICAL TRIAL: NCT07330271
Title: A Multicenter, Randomized Controlled Trial of PTC-Guided Personalized Therapy for Peritoneal Mesothelioma
Brief Title: PTC-Guided Therapy for Peritoneal Mesothelioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other); Cangzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Yan Li, Professor of Oncology and Director of the Department of Peritoneal Oncology, Beijing Tsinghua Chang Gung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25879-0-02
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Peritoneal Mesothelioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: PTC guided individualized treatment
- Control Group (Active Comparator)
  Interventions: Drug: Standard chemotherapy regimens

INTERVENTIONS:
Drug: PTC guided individualized treatment — According to the PTC drug sensitivity test, the types of chemotherapy combined with targeted and immune drugs were determined
  Arms: Experimental Group
Drug: Standard chemotherapy regimens — According to the previous study, the patient received gemcitabine + oxaliplatin + apatinib standard treatment regimen
  Arms: Control Group

SUMMARY:
Official Title: A Study of Key Parameters and Mechanisms in Personalized Diagnosis and Treatment Using Tumor Models

Why is this study being done? This research study is for adults with a type of cancer called Malignant Peritoneal Mesothelioma (MPM). Currently, it is hard for doctors to know which treatment will work best for each patient after surgery. This study will test a new, personalized way to choose treatments using a model grown from a patient's own tumor in the lab, called a Patient-derived tumor-like cell cluster (PTC) model. The main goal is to see if using this PTC model to guide treatment can help patients live longer without their cancer getting worse, compared to a standard chemotherapy treatment.

Who can participate? Adults aged 18 and older with a specific type of MPM (epithelioid or biphasic) who are planned to have surgery and heated chemotherapy (CRS+HIPEC) and can provide a tumor sample for the PTC model may be eligible.

What will happen in the study?

* Participants will be randomly assigned to one of two groups by chance, like flipping a coin.
* Standard Treatment Group: This group will receive the standard chemotherapy combination of Gemcitabine, Oxaliplatin, and Apatinib.
* Personalized Treatment Group: This group will have a PTC model made from their tumor. The model will be tested with different drugs (chemotherapy, targeted therapy, and immunotherapy) in the lab. The treatment that works best on the model will be chosen for the patient.
* Both groups will receive their assigned treatment for 6 cycles.
* Participants will be followed for several years to see how they are doing, through clinic visits and scans.

What are the possible benefits? Participants in the personalized treatment group might receive a therapy that is more effective for their specific cancer. The information from this study may help doctors better treat future patients with MPM.

What are the possible risks? The risks include side effects from cancer treatments, which can include low blood cell counts, nausea, vomiting, high blood pressure, liver problems, and tiredness. There is also a risk that the PTC model may not grow successfully in the lab, or that the drug that works in the model may not work as well in the body. The study team will closely monitor all participants for any side effects and manage them promptly.

Who is paying for the study? This study is funded by the National Key R&D Program of China.

Where is the study taking place? The study is conducted at multiple hospitals in China, including Beijing Tsinghua Changgung Hospital, Beijing Shijitan Hospital, and Cangzhou Central Hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet ALL of the following criteria to be eligible for the study:

* Aged 18 years or older.
* Histopathologically confirmed diagnosis of epithelioid or biphasic malignant peritoneal mesothelioma (MPM).
* Scheduled to undergo cytoreductive surgery (CRS) combined with hyperthermic intraperitoneal chemotherapy (HIPEC) and subsequent adjuvant therapy.
* Availability of sufficient fresh tumor tissue sample obtained during surgery for Patient-derived tumor-like cell clusters (PTC) drug sensitivity testing.
* Karnofsky Performance Status (KPS) score > 60.
* Adequate hematologic function:
* White blood cell count ≥ 3.5 × 10⁹/L
* Platelet count ≥ 80 × 10⁹/L
* Adequate hepatic function:
* Total bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) < 2 × upper limit of normal (ULN)
* Adequate renal function:
* Serum creatinine < 1.2 × ULN
* Adequate cardiac and pulmonary function to tolerate major surgery, as assessed by the investigator.
* Voluntarily agrees to participate by providing written informed consent and demonstrates good compliance.

Exclusion Criteria:

Patients who meet ANY of the following criteria will be excluded from the study:

* Presence of concurrent severe medical comorbidities that, in the investigator's judgment, preclude tolerance to the study treatment.
* Diagnosis of another active malignant tumor during the screening process, which may interfere with the study outcomes.
* Considered by the investigator to be unsuitable for participation in this study for any other reason (e.g., psychological, familial, or social factors).
* Unwillingness to accept the assigned treatment regimen or the required follow-up schedule.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 5 years.

SECONDARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented disease progression or death from any cause, whichever comes first, assessed up to 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Tsinghua University affiliated Beijing Tsinghua Changgung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided